CLINICAL TRIAL: NCT05660681
Title: A Single-Center, Double-Masked, Randomized Study Evaluating the Tolerability and Efficacy of CWT-f-002 Lubricant Eye Drops Compared to Systane® Preservative-Free Eye Drops in the Treatment of the Signs and Symptoms of Dry Eye Disease (DED)
Brief Title: Evaluation of the Tolerability and Efficacy of CWT-f-002 Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calm Water Therapeutics LLC (Industry)
Collaborators: Andover Research Eye Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWT-002
Record Dates: First submitted 2022-11-23; First posted 2022-12-21 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye Disease
Keywords: Corneal Epitheliopathy; Tear Film Stability
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Glycerol; polyethylene glycol 400

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked, single-center, interventional trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- glycerin 0.7%/PEG 400 0.3% (Experimental): 20 patients will receive glycerin 0.7%/PEG 400 0.3% lubricant eye drops three times per day for 28 days.
  Interventions: Drug: glycerin 0.7%/PEG 400 0.3%
- polyethylene glycol 400 0.4%/propylene glycol 0.3% (Active Comparator): 10 patients will receive polyethylene glycol 400 0.4%/propylene glycol 0.3% lubricant eye drops three times per day for 28 days.
  Interventions: Drug: polyethylene glycol 400 0.4%/propylene glycol 0.3%

INTERVENTIONS:
Drug: glycerin 0.7%/PEG 400 0.3% — Eye drop with active agents from the OTC Monograph.
  Other Names: CWT-f-002
  Arms: glycerin 0.7%/PEG 400 0.3%
Drug: polyethylene glycol 400 0.4%/propylene glycol 0.3% — Eye drop with active agents from the OTC Monograph.
  Other Names: Systane (R)
  Arms: polyethylene glycol 400 0.4%/propylene glycol 0.3%

SUMMARY:
The primary objective is to evaluate the tolerability and efficacy of CWT-f-002 lubricant eye drops in the treatment of the signs and symptoms of dry eye disease.

DETAILED DESCRIPTION:
In this study CWT-f-002 lubricant eye drop is being evaluated in subjects with dry eye. This OTC eye drop has previously shown promising results in multiple preclinical and clinical settings. The active comparator for this study is Systane (R). Ingredient lists as follows. CWT-f-002: Active Ingredients are glycerin 0.7% and polyethylene glycol 400 0.4%. Inactive ingredients are mannitol, polylysine-graft-polyethylene glycol, sterile water for injection, and sodium phosphate buffer. Systane: Active ingredients are polyethylene glycol 400 0.4% and propylene glycol 0.3%. Inactive ingredients are boric acid, calcium chloride, hydroxypropyl guar, magnesium chloride, potassium chloride, purified water, sodium chloride, zinc chloride. Systane (R) may contain hydrochloric acid and/or sodium hydroxide to adjust pH. Both products are preservative free and supplied in unit dosers.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have a reported history of dry eye for at least 6 months
* Have a Tear Film Breakup Time (TFBUT) measurement of >1 and <7 seconds at Visit 1

Exclusion Criteria:

* Known contraindications or sensitivities to the use of the study treatment or any of its components
* Have a clinically significant slit lamp finding at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters
* Have a condition (ocular or systemic) that the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Tear Film Break-up Time | 15 minutes after eye drop instillation
  State-of-the-art methodology to assess tear stability.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gomes, MS, Study Director — Andover Research Eye Institute
Locations (1):
- Andover Research Eye Institute, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Farrand KF, Fridman M, Stillman IO, Schaumberg DA. Prevalence of Diagnosed Dry Eye Disease in the United States Among Adults Aged 18 Years and Older. Am J Ophthalmol. 2017 Oct;182:90-98. doi: 10.1016/j.ajo.2017.06.033. Epub 2017 Jul 10. PMID 28705660
- [Background] Gensheimer WG, Kleinman DM, Gonzalez MO, Sobti D, Cooper ER, Smits G, Loxley A, Mitchnick M, Aquavella JV. Novel formulation of glycerin 1% artificial tears extends tear film break-up time compared with Systane lubricant eye drops. J Ocul Pharmacol Ther. 2012 Oct;28(5):473-8. doi: 10.1089/jop.2011.0053. Epub 2012 May 3. PMID 22554205